CLINICAL TRIAL: NCT05267275
Title: Effect of Splenic Flexure Mobilization With Extended Resection of the Proximal Colon for Rectal Cancer With Neoadjuvant Radiotherapy on Postoperative Complications
Brief Title: Extended Resection for Rectal Cancer With Neoadjuvant Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202111-226
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-11

CONDITIONS: the Incidence of Complications Related to Rectal Anastomosis After Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- extended resection with splenic flexure mobilization (Experimental)
  Interventions: Procedure: extended resection with splenic flexure mobilization

INTERVENTIONS:
Procedure: extended resection with splenic flexure mobilization — During the operation, the splenic flexure of the colon was first freed, and then the physiological adhesion site of the sigmoid colon was located. Routine laparoscopic or open rectal cancer radical resection (D3 dissection + high ligation) was performed. The proximal end of the colon is disconnected 10-15cm away from the physiological adhesion site of the sigmoid colon. The anastomosis method was manual anastomosis or stapler anastomosis, and a prophylactic ileal loop ostomy was routinely performed.

SUMMARY:
Preoperative neoadjuvant therapy has become the guideline-recommended standard treatment for patients with locally advanced or mid-to-low rectal cancer with suspected regional lymph node metastasis. However, preoperative neoadjuvant radiotherapy caused radiation damage to the pelvic bowel, resulting in varying degrees of edema, vascular stiffness, and insufficient blood supply. According to the traditional rectal cancer surgery, the proximal bowel resection only needs to be more than 10cm above the upper edge of the tumor. However, this range of resection cannot remove all the damaged proximal bowel, and using the damaged proximal bowel for anastomosis may lead to the risk of anastomotic-related complications (including anastomotic leakage, anastomotic stenosis, and anastomotic proximal bowel stiffness, etc.) also increased. Therefore, extended resection of the proximal bowel with splenic flexure mobilization and using healthy proximal bowel for anastomosis may help reduce the incidence of complications related to rectal anastomosis after neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mid-low rectal cancer who received preoperative neoadjuvant therapy (tumor distance ≤12cm from the anus);
2. The preoperative local stage is cT3-4N0-2M0 or cT3-4N0-2M1 (M1 is limited to liver metastases that can be surgically removed at the same time)
3. Preoperative neoadjuvant therapy (long-course concurrent chemoradiation or TNT)
4. Aged between 18-75 years old;
5. ASA rating: 0-2
6. ECOG Score: 0-2
7. BMI 18-30 kg/m2;
8. Radical surgical resection is expected to be possible on the basis of preserving the anus;
9. Sign the informed consent document.

Exclusion Criteria:

1. History of other malignant tumors;
2. Emergency surgery patients;
3. Severe underlying diseases, unable to tolerate surgery;
4. Without informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
incidence of complications related to rectal anastomosis | From the end of the surgery to 1 year after ileostomy closure

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China